CLINICAL TRIAL: NCT02103309
Title: Comparative Evaluation of Contact Lens Centering of DAILIES® AquaComfort Plus® Versus 1-DAY ACUVUE® MOIST®
Brief Title: Comparative Evaluation of Contact Lens Centering of DAILIES® AquaComfort Plus® Versus 1-DAY ACUVUE® MOIST® in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M-13-050
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Refractive Error; Myopia; Myopic Astigmatism
Keywords: Soft contact lenses; DACP
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DACP, then 1DAM (Other): Nelfilcon A contact lenses worn first, then etafilcon A contact lenses worn second. Each product worn bilaterally (in both eyes) for 1 week in a daily disposable mode.
  Interventions: Device: Nelfilcon A contact lenses; Device: Etafilcon A contact lenses
- 1DAM, then DACP (Other): Etafilcon A contact lenses worn first, then nelfilcon A contact lenses worn second. Each product worn bilaterally (in both eyes) for 1 week in a daily disposable mode.
  Interventions: Device: Nelfilcon A contact lenses; Device: Etafilcon A contact lenses

INTERVENTIONS:
Device: Nelfilcon A contact lenses
  Other Names: DAILIES® AquaComfort® Plus; DACP
Device: Etafilcon A contact lenses
  Other Names: 1-DAY ACUVUE® MOIST®

SUMMARY:
The purpose of this study is to evaluate lens centration and subjective impressions of DAILIES® AquaComfort Plus® (DACP) lenses compared to 1-DAY ACUVUE® MOIST® (1DAM) lenses in ball sports players.

ELIGIBILITY:
Inclusion Criteria:

* Those who can understand the clinical study objectives and provide written informed consent. Legal representative or parental consent required if under age 20
* Those who regularly wear soft contact lenses in both eyes for a minimum of 8 hours per day and 5 days per week
* Those who play ball sports at least 1 day per week
* Those who need vision correction because of myopia or mild myopic astigmatism, who are eligible for use of the study device, and who can attain a visual acuity of at least 1.0 with correction
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Those who regularly wear the study device
* Those who require ocular treatment with eye drops
* Those who have a condition contraindicating soft contact lens wear, such as eye irritation
* Those who have had ocular disorder or ocular surgery that may affect soft contact lens wear within 3 months before the start of the study
* Those who are participating in another clinical study or research or have a plan of such participation during the present study
* Women who are pregnant or intend to become pregnant during the study
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L. Zoota, MPH, CCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 study centers located in Japan.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | DACP, Then 1DAM | 1DAM, Then DACP
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Groups:
- Overall: DAILIES® AquaComfort Plus® and 1-Day ACUVUE® MOIST® contact lenses worn in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Investigator-Rated Lens Centration
Description: Lens centration was assessed by the investigator using slit-lamp microscopy and rated on a 5-point scale, where 0=Optimal and 4=Severe decentration. Both eyes contributed to the mean.
Time Frame: After 1 week of wear
Population: This analysis population includes all enrolled participants minus missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DACP: Nelfilcon A contact lenses worn bilaterally (in both eyes) for 1 week in a daily disposable mode.
- 1DAM: Etafilcon A contact lenses worn bilaterally (in both eyes) for 1 week in a daily disposable mode.
Arm/Group | DACP | 1DAM
Number analyzed (Participants) | 41 | 39
units on a scale | 0.34 (0.47) | 0.73 (0.83)

2. Secondary Outcome: Mean Investigator-Rated Lens Fit
Description: Lens fit was assessed by the investigator and rated on a 5-point scale with -2=Unacceptable tight fit, -1=Acceptable tight fit, 0=Optimal, 1=Acceptable loose fit, and 2=Uacceptable loose fit. Both eyes contributed to the mean.
Time Frame: After 1 week of wear
Population: This analysis population includes all enrolled participants minus missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DACP | 1DAM
Number analyzed (Participants) | 41 | 39
units on a scale | 0.24 (0.42) | 0.28 (0.50)

3. Secondary Outcome: Average Subjective Ratings Score (Lens Handling and Overall Vision)
Description: The participant rated the handling and overall vision of the contact lenses on a 10-point scale, where 10=Excellent and 1=Poor. Both eyes contributed to the mean.
Time Frame: After 1 week of wear
Population: This analysis population includes all enrolled participants minus missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DACP | 1DAM
Number analyzed (Participants) | 42 | 42
units on a scale
  Ease of insertion | 7.8 (2.0) | 6.4 (2.7)
  Ease of removal | 7.2 (2.5) | 8.2 (1.9)
  Overall vision | 8.1 (1.9) | 7.4 (2.2)

4. Secondary Outcome: Average Subjective Ratings Score (Lens Wearing Conditions and Visual Performance During Ball Sports)
Description: The participant rated the lens wearing conditions and visual performance of the contact lenses during ball sports on a 10-point scale, where 10=Agree and 1=Disagree. "Overall Vision" was rated with 10=Excellent and 1=Poor. Both eyes contributed to the mean.
Time Frame: After 1 week of wear
Population: This analysis population includes all enrolled participants minus missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DACP | 1DAM
Number analyzed (Participants) | 42 | 42
units on a scale
  Sense of discomfort | 3.5 (2.6) | 3.8 (2.6)
  A lens comes off my eye | 2.4 (2.2) | 2.5 (2.2)
  A lens becomes out of place | 3.3 (2.5) | 4.0 (2.9)
  Improves my vision/widens my vision | 6.3 (2.4) | 5.8 (2.4)
  My vision does not become blurry | 6.3 (2.5) | 6.0 (2.5)
  Do not lose a sense of perspective/distance | 6.8 (3.3) | 6.4 (2.2)
  Does not give me improper vision | 7.4 (2.2) | 7.1 (2.3)
  Enables me to see clearly at important occasion | 6.9 (2.4) | 6.5 (2.2)
  Improves my vision when playing sports | 6.6 (2.5) | 6.3 (2.0)
  Overall vision | 7.2 (2.1) | 7.1 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (1 month). This analysis group includes (Safety Population). based on treatment-specific exposure
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in patients, users or other persons, whether or not related to the medical device.
Arm/Group | DACP | 1DAM
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.